CLINICAL TRIAL: NCT02656953
Title: The Impact of Wearing VDU Lenses Versus Progressive Lenses on Musculoskeletal and Visual Complaints in VDU Workers With Work Related Neck Complaints: A Randomized Controlled Trial
Brief Title: The Impact of Lenses on Musculoskeletal and Visual Complaints in VDU Workers With Neck Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20150115
Record Dates: First submitted 2015-12-18; First posted 2016-01-15 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Neck Pain
Keywords: VDU workers; VDU lenses; Neck complaints; Visual complaints
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VDU lenses (Experimental): VDU lenses provide a clear vision of the intermediate zone at a distance of approximately 70 centimeters, which is closer than distant vision at a distance of more than 2 meters (e.g. driving), but further than near vision at a distance of 40 centimeters (e.g. reading), so the computer screen is seen clear without the need for excessive focusing effort or bad postures. In this study Zeiss® Officelens Plus lenses with a Silhouette® frame were used.
  Interventions: Other: VDU lenses (Zeiss® Officelens Plus)
- Progressive lenses (Active Comparator): Progressive lenses or multifocal lenses provide a continuous range of focal power between near and far distances.Progressive lenses have some lens power for the intermediate zone as well, but this zone might not be large enough for comfortable and ergonomic computer work. In this study Zeiss® Multifocal Precision Plus lenses with a Silhouette® frame were used.
  Interventions: Other: Progressive lenses (Zeiss® Multifocal Precision Plus)

INTERVENTIONS:
Other: VDU lenses (Zeiss® Officelens Plus) — The treatment group (n=22) was given progressive VDU glasses (Zeiss® Officelens Plus), specially designed for VDU work. The participants were asked to wear their new glasses for six months during computer work.
  Arms: VDU lenses
Other: Progressive lenses (Zeiss® Multifocal Precision Plus) — The comparison group (n=18) was given progressive glasses (Zeiss® Multifocal Precision Plus). The participants were asked to wear their new glasses for six months during computer work.
  Arms: Progressive lenses

SUMMARY:
The aim of this study is to investigate the impact of wearing visual display units (VDU) lenses versus progressive lenses on musculoskeletal and visual complaints in VDU workers with work related neck complaints. This will be evaluated by means of questionnaires (Neck Disability Index and Visual Fatigue Questionnaire), muscle tone, elasticity and stiffness, pressure pain threshold and 2D video analysis of head posture during a VDU task.

DETAILED DESCRIPTION:
The use of visual display units (VDU) is often accompanied by physical complaints of the neck, shoulder, forearm and hand, especially in people who make extensive use of computers at work. Besides this, VDU operators also experience eye discomfort and vision problems when working with the computer for a long period.

With the increase of computer use, VDU glasses were developed. They provide a clear vision of the intermediate zone at a distance of approximately 70 centimeters, which is closer than distant vision at a distance of more than 2 meters (e.g. driving), but further than near vision at a distance of 40 centimeters (e.g. reading), so the computer screen is seen clear without the need for excessive focusing effort or bad postures. Progressive lenses have some lens power for this intermediate zone as well, but this zone might not be large enough for comfortable and ergonomic computer work. VDU glasses are often progressive glasses as well, so they can be used to read and see things beyond the computer screen clear during computer work.

The research question of this study is "What is the impact of wearing progressive VDU lenses versus progressive lenses, for six months, on both musculoskeletal and visual complaints in VDU workers with work related neck complaints ?"

To find an answer to this question, 40 VDU workers (men and women) with work related neck/shoulder complaints, were recruited from a bank office where they perform predominantly VDU work. All participants will receive information and have to sign an informed consent form.

A questionnaire concerning visual and musculoskeletal complaints, in which the Neck Disability Index (NDI) Questionnaire had to be completed at the beginning of the experiment. Participants were tested with their old glasses in a landscape office while performing a 20 minute VDU task. Before and after the task, viscoelastic properties (MyotonPRO®) of the trapezius muscle and the PPT (WagnerTM FDX 50 hand-held pressure algometer) of the trapezius muscle, the levator scapulae muscle and the infraspinatus muscle were measured. A 2D video analysis was performed during the task.The Forward Head Angle (FHA) and the Forward Shoulder Angle (FSA) was measured afterwards. After this, participants were asked to fill out a short questionnaire, in which the Visual Fatigue Questionnaire was included, every two weeks during two months. On the 15th of June, 2015 the participants received new glasses and were asked to wear these for six months during computer work. During this period the same short questionnaire had to be filled out every two weeks. The test procedure will be repeated with the new glasses after six months of wearing these. A shorter version of the first questionnaire will be completed at the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 4 hours a day and 20 hours a week of VDU work
* Work related neck/shoulder complaints
* Difference in spectacle correction for presbyopia and myopia of minimum 1.5 dioptres

Exclusion Criteria:

* Active eye disease that can't be corrected with eyeglasses
* Drugs that strongly influence eye or muscle function

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in functionality using the Neck disability index (NDI) | At baseline and six months
  The NDI consists of ten questions concerning pain and daily living activities such as lifting, reading, driving, etc. and the maximum score is 50.
Change in visual complaints using the Visual Fatigue Questionnaire | At baseline and six months
  The questionnaire consists of 15 questions which have to be answered on a visual analogue scale ranging from zero to ten. It enquires eye strain, impaired vision, impaired eye surface and problems of the outside of the eyes, headache for example. The maximum score is 10.

SECONDARY OUTCOMES:
Change in muscle elasticity by using the MyotonPRO® device | At baseline and six months
  The MyotonPRO® is a digital device that measures the elasticity (logarithmic decrement) of a muscle.
Change in muscle stiffness by using the MyotonPRO® device | At baseline and six months
  The MyotonPRO® is a digital device that measures muscle stiffness, this is expressed in N/m.
Change in muscle tone by using the MyotonPRO® device | At baseline and six months
  The MyotonPRO® is a digital device that measures muscle tone, this is expressed in Hz
Change in pressure pain threshold by using the WagnerTM FDX 50 hand-held pressure algometer | At baseline and six months
  The WagnerTM FDX 50 hand-held pressure algometer is a digital device that measures the point at which pressure (N) becomes unpleasant, also known as the pressure pain threshold (PPT).
Change in head posture during a VDU task by means of 2D video analysis | At baseline and six months
  A 2D video analysis of the head posture was performed during a VDU task using a Logitech® webcam with a Zeiss® Tessar HD 1080p lens and MaxTRAQ and MaxMATE software.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, PhD, Principal Investigator — University Ghent

IPD SHARING:
Plan to Share IPD: No